CLINICAL TRIAL: NCT05865340
Title: To Exam the Efficacy of Oral Health and Mediterranean Diet Interventions in Preventing Cognitive Decline Among Older Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-12-013BCF
Record Dates: First submitted 2023-04-05; First posted 2023-05-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment (MCI); Oral Health; Mediterranean Diet
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Oral Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- oral health + MED diet (Other): oral health + MED diet education
  Interventions: Behavioral: oral health + MED diet
- oral health (Other): oral health education
  Interventions: Behavioral: oral health
- MED diet (Other): MED diet education
  Interventions: Behavioral: MED diet
- compare (No Intervention)

INTERVENTIONS:
Behavioral: oral health + MED diet — oral health + MED diet education
  Arms: oral health + MED diet
Behavioral: oral health — oral health education
  Arms: oral health
Behavioral: MED diet — MED diet education
  Arms: MED diet

SUMMARY:
At present, many literatures have confirmed that the Mediterranean diet has the effect of delaying cognitive degeneration in patients with mild cognitive impairment, and can also slow down the speed of brain atrophy. In addition to the highly respected Mediterranean diet every year, several years of foreign research have found The maintenance of oral hygiene also has a significant relationship with the decline of cognitive function. The intervention of "oral hygiene" is a new intervention method that has started in recent years. Oral health will affect the overall health status, physical function, diet and nutritional status of the elderly. In particular, older adults with poor oral health are more likely to suffer from mild cognitive impairment. The relationship between oral health and nutrition and overall health is inseparable. If the concept of healthy eating (Mediterranean diet) recognized by the public is used and oral health education is involved at the same time. To allow patients with mild cognitive impairment to maintain oral health care in daily life, and to increase the knowledge of the Mediterranean diet and try to follow the rules of the Mediterranean diet, whether there is a more significant impact on these patients.

DETAILED DESCRIPTION:
This trial is expected to enroll 120 subjects, which will be accepted by the relevant researchers who carry out this study. In the pre-test part, all subjects will receive the Montreal Intelligence Test (MoCA) and Mini Intelligence Examination (MMSE) and collect MEDAS-14 Item, Oral Health Assessment Tool, OHAT and evaluation data of Taiwan Frailty Criteria of Taiwan. After completing the 12-week oral health and Mediterranean diet education intervention, all subjects will undergo post-test follow-up evaluation (MoCA, MMSE, MEDAS-14 item, OHAT and Frailty Criteria), and all subjects will be assessed 12 weeks after the intervention The subjects were followed up with follow-up cognitive function tracking (MoCA, MMSE, MEDAS-14 item, OHAT and Frailty Criteria). Finally, all the data were statistically analyzed to study which of the individual measures and the combined measures had a more significant cognitive effect on MCI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Over or equal to 50 years old
2. CDR score is less than or equal to 0.5 or MMSE score is 24-30 (including 24 and 30)
3. Conscious/complaint of cognitive decline

Exclusion Criteria:

1. Dementia
2. Acute and significant mental illness in the past three months
3. Acute serious medical and surgical diseases in the past three months
4. Symptoms of delusions, hallucinations or delirium in the past three months
5. Severe visual and hearing impairment in the past three months
6. Other conditions that make the patient unable to cooperate: such as not being suitable after screening, not signing the subject's consent form.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
cognitive | 6 months
  MoCA&MMSE
diet | 6 months
  MEDAS-14 item
oral health | 6 months
  OHAT
frailty | 6 months
  Frailty Criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No